CLINICAL TRIAL: NCT01144871
Title: Parental Knowledge and Attitudes of Confidential STI Services for Teens
Brief Title: Parental Knowledge and Attitudes of Confidential Sexually Transmitted Infections (STI) Services for Teens
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: H1095-31348; R01HD053408-01A2 (NIH)
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Sexually Transmitted Infections
Keywords: adolescent; reproductive health; parents; STIs; confidentiality; Examine parental knowledge/attitudes of confidential health services/STI care for adolescents.; Examine how parental knowledge/attitudes affects parent's behavioral intentions to support adolescent's access to confidential care.; Identify key mechanisms to form an intervention to parents knowledge/skills to facilitate teen's access to confidential STI services.
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Male Parent/Guardians: Male Parent/Guardian of Adolescent 12-17 yo. Health care members of either San Francisco General Hospital or Kaiser Permanente Northern California.
- Female Parent/Guardian: Female Parent/Guardian of Adolescent 12-17 yo. Health care members of either San Francisco General Hospital or Kaiser Permanente Northern California.

SUMMARY:
This study will provide new and important information regarding parental knowledge and attitudes of confidential STI and related health care services (prevention, diagnosis and treatment) for teens that may be needed to address the STI epidemic. Using both qualitative and quantitative methods, this study will gather information necessary to develop effective interventions aimed at the often neglected parent component of the teen-parent-health care provider partnership by giving parents knowledge and skills to help them facilitate their adolescent's access to confidential STI services as needed.

DETAILED DESCRIPTION:
Teens' access to confidential services for sexually transmitted infections (STI's) has been assured over time by privacy protections established through statutory and policy routes. Yet, the STI epidemic among youth persists, in part , because many STI's are largely asymptomatic, remain undetected and continue to be transmitted unknowingly. Also, many teens are reluctant to obtain STI services due to embarrassment, fear of disclosure, lack of knowledge about STI diagnosis/treatment, and confidential STI services. How do we bridge the gap between availability and apparent lack of utilization by teens in need of confidential services to prevent STI's and their long term sequelae? One strategy that has been overlooked is the engagement of parents in a partnership with the teen and the provider to effectively guide the developing adolescent towards becoming a responsible and confident adult consumer of health services, especially regarding STI prevention and care including confidential services. Before developing the parental component to a broad-based effort aimed at decreasing the STI rate, especially C. trachomatis, it is important to examine parental knowledge and attitudes towards confidential STI health services for teens and how these might influence parental intention to facilitate their adolescent's accessing appropriate preventive care for STIs. We propose a multi-method research design in 2 phases. Phase 1 comprises a qualitative format (focus groups and 1:1 semi-structured interviews) designed to yield data on parental knowledge and attitudes about confidential STI related health care services for teens. Findings from Phase 1 will then inform Phase 2, a quantitative cross-sectional survey of a random sample of ethnically diverse parents of 12-17 yo teens designed to examine the following questions. First, how does parental knowledge and attitudes about STI confidential care for teens vary according: (a) the adolescent's age and gender; and (b) the specific parental characteristics, e.g., gender, race/ethnicity, insurance status, education, religiosity. Secondly, how does parental knowledge and attitudes about confidential care for teens affect parental behavioral intentions to facilitate their teen's gaining knowledge and skills to be able to access STI preventive confidential services. This research would inform investigations how to strengthen the role of parents and encourage partnerships between health care providers and parents to ultimately improve the health outcomes for teens.

Hypotheses:

1. Parental knowledge of confidential care for adolescents will increase parental intention to facilitate confidential care
2. Parental knowledge of STI's will be positively associated with their perceptions of their teen's susceptibility to/ severity of STI
3. Parental knowledge or suspicion that their adolescent is having sex will be associated with perceptions that their teen is susceptibility to STIs
4. Parental knowledge of STI's and/or knowledge/ suspicion adolescent is having sex will be associated with parental intention to facilitate confidential care
5. Perceived susceptibility/severity of their teen to STI will be associated with a greater intention to facilitate confidential care
6. Perceived benefits of confidential care will be associated with an greater intention to facilitate confidential care
7. Perceived risks/barriers to confidential care (e.g., logistical/billing; busy practice, no policy/time for provider to see teen alone; perceived increase risky teen behavior due to such sexual health discussions) will be negatively associated with intention to facilitate confidential care
8. Perceived self-efficacy will be associated with an greater intention to facilitate confidential care
9. Past behavior/experiences regarding confidential care for parent and/or adolescent will be associated with intention to facilitate confidential care

Specific Aims:

i. To examine parental knowledge and attitudes of confidential health services related to STI care for adolescents

1. To examine how parental knowledge and attitudes of confidentiality regarding STI and related health care services vary according to parent characteristics
2. To examine how parental knowledge and attitudes of confidentiality regarding STI and related health care services vary according to child characteristics

ii. To examine how parental knowledge and attitudes toward confidential STI care affects the parent's behavioral intentions to support their adolescent's access to confidential care

iii. To identify key mechanisms that will form the basis of an intervention to improve parent-health care provider partnerships by giving parents knowledge and skills to help them facilitate their adolescent's access to confidential STI services as needed

ELIGIBILITY:
Inclusion Criteria:

* Parents/Guardians who have adolescents between 12-17 years of age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parents/Guardians who have adolescents between 12-17 years of age
Sampling Method: Non-Probability Sample
Enrollment: 1216 (Actual)
Dates: Start 2007-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Determining parental attitudes regarding confidential health services for their teens | 4 years
  Parental attitudes and knowledge regarding confidential health services will be assessed with focus groups, interviews and phone surveying.

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ann Shafer, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Mission Neighborhood Health Center, San Francisco, California
  - San Francisco General Hospital, San Francisco, California
  - Kaiser Permanente Northern California, San Francisco, California